CLINICAL TRIAL: NCT03490604
Title: Ambulatory Measurement of Physical Activity in Pancreatic Cancer Patients
Acronym: ARABICA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: DROUILLARD AOI 2017
Record Dates: First submitted 2018-03-30; First posted 2018-04-06 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Unresectable Pancreatic Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: wrist-worn accelerometer — accelerometer worn on the patient's wrist, changed every 15 ± 7 days for 6 months when the patient comes for a chemotherapy session
Other: Auto-questionnaires — Questionnaire regarding physical activity over the previous 7 days, questionnaires EORTC QLQ-C30 and EORTC QLQ-PAN26

SUMMARY:
Pancreatic cancer is the 5th leading cause of death from cancer in France. When chemotherapy can be proposed, the choice of treatment is currently based on the patient's profile and expected tolerance. The endpoints currently used in trials, such as time to therapeutic failure, do not take into account the patient's experience of the disease. The use of quality of life questionnaires is often proposed, but frequent missing data and filling time can be a problem. In oncology, some studies have demonstrated, through questionnaires, the link between physical activity and quality of life. In this situation, ambulatory measurement of physical activity by wrist actimetry could be an integrative reflection of the impact of the disease and treatment (efficacy, tolerance) on patients. This type of evaluation, if accepted by patients, could usefully complement the measurement of quality of life in this population. No study has specifically looked at the use of devices of this type in the context of digestive cancer. The investigators propose to evaluate the acceptance of this type of device by pancreatic cancer patients receiving chemotherapy before evaluating its potential interest.

ELIGIBILITY:
Inclusion Criteria:

* Patient with unresectable pancreatic adenocarcinoma for whom an indication for chemotherapy has been decided upon after a multidisciplinary consultation meeting;
* Adult patient;
* Patients able to understand spoken and written French,
* Patient has given consent.

Exclusion Criteria:

* WHO ECOG stage III or IV ;
* Patient suffering from a major physical disability (hemiplegia, paraplegia, myopathy, amputation of a limb);
* Any alteration of comprehension capacities making self-evaluation impossible;
* Protected adult;
* Patient not affiliated to a national health insurance scheme;
* Pregnant or nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients followed in the hospital unit
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
average time wearing the accelerometer, in hours | every 2 weeks for 6 months
  the amount of time the accelerometer is not worn will be estimated using the standard deviation and range of acceleration in each of the 3 axes, calculated for consecutive 15-minute windows

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France